CLINICAL TRIAL: NCT00870077
Title: Effect of a Whey Protein Supplementation on Intrahepatic Lipids in Obese Patients With Non-alcoholic Fatty Liver Disease
Brief Title: A Pilot Study on Whey Protein Supplementation in Non Alcoholic Fatty Liver Disease
Acronym: PROTOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, professor of physiology, University of Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protobese
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Non-alcoholic Fatty Liver Disease; Obesity
Keywords: Intrahepatic fat; obesity; body fat; impaired glucose tolerance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Dietary Supplement: ProWHEY 94 CFM, SponserR

INTERVENTIONS:
Dietary Supplement: ProWHEY 94 CFM, SponserR — 3 times 20g per day

SUMMARY:
An increase in dietary protein intake has been shown to blunt the increase in intrahepatic fat induced by high fat feeding in healthy individuals. The purpose of this study is to determine if a protein supplementation decreases intrahepatic fat in obese patients with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
12 obese patients will be be treated with a dietary whey protein supplementation over 4 weeks. Their intrahepatic fat content, glucose tolerance, and body weight will be evaluated before and after 4 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* BMI higher than 35 kg/m2
* age 18-50 years
* sex male or female
* ASAT/ALAT > 1.8

Exclusion Criteria:

* treatment with hypolemic or antidiabetic agents
* blood glucose > 7 mmol/l
* alcohol intake > 20g/day
* creatinin > 120 umol/l)
* contra-indications to Magnetic resonnance imaging

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
intrahepatic fat | before and after 4 weeks of whey protein supplementation

SECONDARY OUTCOMES:
glucose metabolism | 4-hour oral glucose tolerance test with indirect calorimetry
body weight and body fat | before and after 4 weeks whey protein supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre d'investigations cliniques "cardiomet"/ CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Bortolotti M, Maiolo E, Corazza M, Van Dijke E, Schneiter P, Boss A, Carrel G, Giusti V, Le KA, Quo Chong DG, Buehler T, Kreis R, Boesch C, Tappy L. Effects of a whey protein supplementation on intrahepatocellular lipids in obese female patients. Clin Nutr. 2011 Aug;30(4):494-8. doi: 10.1016/j.clnu.2011.01.006. Epub 2011 Feb 1. PMID 21288612